CLINICAL TRIAL: NCT02961556
Title: General Clinical Study of AJG555 in Pediatric Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJG555/CT2
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Chronic Constipation
Keywords: AJG555; Constipation; Phase 3; Pediatric participants
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AJG555 (Experimental): After 2 weeks of the screening period, participants will be administered AJG555 starting on the day of the formal enrollment and continuing for 12 weeks.
  Interventions: Drug: AJG555

INTERVENTIONS:
Drug: AJG555 — Participants will receive 1 to 6 sachets daily per participants' age and conditions.

SUMMARY:
This baseline-controlled, open-label, multicenter study evaluates the efficacy and safety of AJG555 orally administered for 2 weeks in pediatric participants with chronic constipation. The safety and efficacy of 12 weeks of administration will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

* Participants with chronic constipation
* Age: 2 years old or older and 14 years old or younger (at the time of the informed consent)
* Gender: N/A

Exclusion Criteria:

Main Exclusion Criteria:

* Participants with organic constipation or participants suspected of having organic constipation
* Participants with symptomatic constipation or participants suspected of having symptomatic constipation
* Participants with drug-induced constipation or participants suspected of having drug-induced constipation

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Change from the second week of the screening period in the number of spontaneous bowel movements (SBMs) at the second week of the administration period | Screening; Week 2 of administration period

SECONDARY OUTCOMES:
Change from the second week of the screening period in the number of SBMs at each week of the administration period | Screening; up to Week 12 of administration period
Change from the second week of the screening period in the number of complete SBMs (CSBMs) at each week of the administration period | Screening; up to Week 12 of administration period
Change from the screening period in the number of SBMs at two weeks after the initiation of the administration | Screening; Week 2
Change from the screening period in the number of CSBMs at two weeks after the initiation of the administration | Screening; Week 2 of administration period
Number of days until SBM and CSBM | up to Week 12 of administration period
Change from the second week of the screening period in the total number of SBMs at each week of the administration period | Screening; up to Week 12 of administration period
Percentage of responders for SBM and CSBM at each week of the administration period | up to Week 12 of administration period
Stool consistency measured by the Bristol stool form scale | up to Week 12 of administration period
Usage of rescue medication | up to Week 12 of administration period
Number of pouches of AJG555 administered | up to Week 12 of administration period
Duration of administration of AJG555 | up to Week 12 of administration period

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - EA Pharma Trial Site #1, Yokohama, Kanagawa
  - EA Pharma Trial Site #2, Yokohama, Kanagawa
  - EA Pharma Trial Site #1, Bunkyo, Tokyo
  - EA Pharma Trial Site #1, Hutyu, Tokyo
  - EA Pharma Trial Site #1, Ōta-ku, Tokyo
  - EA Pharma Trial Site #1, Setagaya City, Tokyo
  - EA Pharma Trial Site #2, Setagaya City, Tokyo
  - EA Pharma Trial Site #1, Shinjuku, Tokyo
  - EA Pharma Trial Site #2, Shinjuku, Tokyo
  - EA Pharma Trial Site #1, Hiroshima
  - EA Pharma Trial Site #1, Saitama